CLINICAL TRIAL: NCT01424150
Title: Restrictive Versus Liberal Fluid Therapy in Major Abdominal Surgery
Brief Title: REstrictive Versus LIbEral Fluid Therapy in Major Abdominal Surgery: RELIEF Study
Acronym: RELIEF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayside Health (Other Government)
Collaborators: National Health and Medical Research Council, Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 164/11 Pilot - 544/12 Main
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Results first posted 2025-01-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2017-08

CONDITIONS: Abdominal Surgery
Keywords: Postoperative fluid; surgery; anaesthesia; fluid; mortality; morbidity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liberal (Experimental): At the commencement of surgery a bolus of Hartmann's balanced salt crystalloid 10 ml/kg followed by 8 ml/kg/h will be administered until the end of surgery. A maintenance infusion will then continue at 1.5 ml/kg/h, for at least 24 hours, but this can be reduced postoperatively if there is evidence of fluid overload and no hypotension, and increased if there is evidence of hypovolaemia or hypotension. Alternative fluid types (crystalloid, dextrose, colloid) and electrolyte supplements will be allowed postoperatively in order to account for local preferences and patient biochemistry, for which we will collect data.
  Interventions: Other: Liberal fluid therapy
- Restrictive (Experimental): Will provide less than 2.0 L water and 120 mmol sodium per day. Induction of anaesthesia will limit IV bolus fluid to ≤5 ml/kg; no other IV fluids will be used at the commencement of surgery (unless indicated by goal-directed device [see below]). Hartmann's balanced salt crystalloid 5 ml/kg/h will be administered until the end of surgery, and bolus colloid/blood used intraoperatively to replace blood loss (ml for ml); then an infusion at 1 ml/kg/h until expedited cessation of IV fluid therapy within 24 hours. The rate of postoperative fluid replacement can be reduced if there is evidence of fluid overload and no hypotension, and can be increased if there is hypotension AND evidence of hypovolaemia.
  Interventions: Other: Restrictive fluid therapy

INTERVENTIONS:
Other: Liberal fluid therapy — Liberal protocol group is designed to provide approximately 6.0L per day.
  Arms: Liberal
Other: Restrictive fluid therapy — Restrictive protocol group is designed to provide less than 2.0 L water and 120 mmol sodium per day.
  Arms: Restrictive

SUMMARY:
The optimal fluid regimen, haemodynamic (or other) targets and fluid choice (colloid or crystalloid) for patients undergoing major surgery are based on rationales that are not supported by strong evidence. Practices vary substantially, guidelines are vague, small trials and meta-analyses are contradictory. The strongest and most consistent evidence, and biological plausibility because of tissue edema, supports a restrictive fluid strategy. But other evidence supports goal-directed therapy, requiring additional IV fluid. There is no good evidence that use and choice of colloids improves outcome. RELIEF will study the effects of fluid restriction, and the possible effect-modification of goal-directed therapy and colloids. The first will be randomly assigned; the latter will be measured covariates dictated by local practices and beliefs.

Study Hypotheses A restrictive fluid regimen for adults undergoing major abdominal surgery leads to reduced complications and improved disability-free survival when compared with a liberal fluid regimen.

Secondary hypothesis: The effects of fluid restriction are similar whether or not goal-directed therapy is used (assessed as a statistical test of interaction). A restrictive fluid regimen will reduce a composite of 30-day septic complications and mortality.

DETAILED DESCRIPTION:
The investigators have completed a pilot study of 82 subjects to test the feasibility of the trial (2011), and are currently doing a cost-effectiveness substudy (2012-13)

1. AIM OF THE TRIAL To investigate the effectiveness of fluid restriction (vs. liberal), and the possible effect-modification of goal-directed therapy (eg. oesophageal Doppler, Flotrac®). The first will be randomly assigned; the latter will be measured covariates according to local practices and beliefs.

The optimal fluid regimen and haemodynamic (or other) targets for patients undergoing major surgery are based on rationales that are not supported by strong evidence. Practices vary substantially; guidelines are vague, small trials and meta-analyses are contradictory. The strongest and most consistent evidence, and biological plausability regarding tissue oedema, supports a restrictive fluid strategy. There is less (and more contradictory) evidence supporting goal-directed therapy using a flow-directed device and/or dopexamine, and use and choice of colloids. A large, definitive clinical trial evaluating perioperative fluid replacement in major surgery is required.

Study Hypotheses A restrictive fluid regimen for adults undergoing major abdominal surgery leads to reduced complications and improved disability-free survival when compared with a liberal fluid regimen.

Secondary hypotheses: The effects of fluid restriction are similar whether or not goal-directed therapy is used (assessed as a statistical test of interaction). A restrictive fluid regimen will reduce a composite of 30-day septic complications and mortality.

ELIGIBILITY:
Inclusion criteria:

1. Adults (≥18 years) undergoing elective major surgery and providing informed consent
2. All types of open or lap-assisted abdominal or pelvic surgery with an expected duration of at least 2 hours, and an expected hospital stay of at least 3 days (for example, oesophagectomy, gastrectomy, pancreatectomy, colectomy, aortic or aorto-femoral vascular surgery, nephrectomy, cystectomy, open prostatectomy, radical hysterectomy, and abdominal incisional hernia repair)
3. At increased risk of postoperative complications, defined as at least one of the following criteria:

   * age ≥70 years
   * known or documented history of coronary artery disease
   * known or documented history of heart failure
   * diabetes currently treated with an oral hypoglycaemic agent and/or insulin
   * preoperative serum creatinine >200 µmol/L (>2.8 mg/dl)
   * morbid obesity (BMI ≥35 kg/m²)
   * preoperative serum albumin <30 g/L
   * anaerobic threshold (if done) <12 mL/kg/min
   * or two or more of the following risk factors:

     * ASA 3 or 4
     * chronic respiratory disease
     * obesity (BMI 30-35 kg/m²)
     * aortic or peripheral vascular disease
     * preoperative haemoglobin <100 g/L
     * preoperative serum creatinine 150-199 µmol/L (>1.7 mg/dl)
     * anaerobic threshold (if done) 12-14 mL/kg/min

Exclusion Criteria

1. Urgent or time-critical surgery
2. ASA physical status 5 - such patients are not expected to survive with or without surgery, and their underlying illness is expected to have an overwhelming effect on outcome (irrespective of fluid therapy)
3. Chronic renal failure requiring dialysis
4. Pulmonary or cardiac surgery - different pathophysiology, and thoracic surgery typically have strict fluid restrictions
5. Liver resection - most units have strict fluid/CVP limits in place and won't allow randomisation
6. Minor or intermediate surgery, such as laparoscopic cholecystectomy, transurethral resection of the prostate, inguinal hernia repair, splenectomy, closure of colostomy - each of these are typically "minor" surgery with minimal IV fluid requirements, generally low rates of complications and mostly very good survival.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul S Myles, MB.BS, MPH, MD, FANZCA, Study Chair — Alfred Hospital, Monash University
Locations (1):
- Alfred Hospital, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bihari S, Dixon DL, Painter T, Myles P, Bersten AD. Understanding Restrictive Versus Liberal Fluid Therapy for Major Abdominal Surgery Trial Results: Did Liberal Fluids Associate With Increased Endothelial Injury Markers? Crit Care Explor. 2021 Jan 25;3(1):e0316. doi: 10.1097/CCE.0000000000000316. eCollection 2021 Jan. PMID 33521643
- [Derived] Gurunathan U, Rapchuk IL, Dickfos M, Larsen P, Forbes A, Martin C, Leslie K, Myles PS. Association of Obesity With Septic Complications After Major Abdominal Surgery: A Secondary Analysis of the RELIEF Randomized Clinical Trial. JAMA Netw Open. 2019 Nov 1;2(11):e1916345. doi: 10.1001/jamanetworkopen.2019.16345. PMID 31774526
- [Derived] Myles PS, McIlroy DR, Bellomo R, Wallace S. Importance of intraoperative oliguria during major abdominal surgery: findings of the Restrictive versus Liberal Fluid Therapy in Major Abdominal Surgery trial. Br J Anaesth. 2019 Jun;122(6):726-733. doi: 10.1016/j.bja.2019.01.010. Epub 2019 Feb 16. PMID 30916001
- [Derived] Myles PS, Bellomo R, Corcoran T, Forbes A, Peyton P, Story D, Christophi C, Leslie K, McGuinness S, Parke R, Serpell J, Chan MTV, Painter T, McCluskey S, Minto G, Wallace S; Australian and New Zealand College of Anaesthetists Clinical Trials Network and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus Liberal Fluid Therapy for Major Abdominal Surgery. N Engl J Med. 2018 Jun 14;378(24):2263-2274. doi: 10.1056/NEJMoa1801601. Epub 2018 May 9. PMID 29742967
- [Derived] Myles P, Bellomo R, Corcoran T, Forbes A, Wallace S, Peyton P, Christophi C, Story D, Leslie K, Serpell J, McGuinness S, Parke R; Australian and New Zealand College of Anaesthetists Clinical Trials Network, and the Australian and New Zealand Intensive Care Society Clinical Trials Group. Restrictive versus liberal fluid therapy in major abdominal surgery (RELIEF): rationale and design for a multicentre randomised trial. BMJ Open. 2017 Mar 3;7(3):e015358. doi: 10.1136/bmjopen-2016-015358. PMID 28259855

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Liberal | Restrictive
Started | 1501 | 1499
Completed | 1493 | 1490
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Population: 2983 (99.4%) met the inclusion criteria for the modified intention-to treat population (1490 in the restrictive fluid group and 1493 in the liberal fluid group)
Groups:
- Total: Total of all reporting groups
Arm/Group | Liberal | Restrictive | Total
Number analyzed (Participants) | 1493 | 1490 | 2983
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (13) | 66 (13) | 66 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 710 | 719 | 1429
  Male | 783 | 771 | 1554
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 841 | 836 | 1677
  Canada | 247 | 250 | 497
  United Kingdom | 134 | 141 | 275
  Hong Kong | 116 | 111 | 227
  United States | 75 | 74 | 149
  New Zealand | 48 | 46 | 94
  Italy | 32 | 32 | 64
American Society Anesthesiologists (ASA) Physical Status [Count of Participants; unit: Participants] — The ASA physical status classification system is a system for assessing the fitness of patients before surgery. In 1963 the American Society of Anesthesiologists (ASA) adopted the five-category physical status classification system; a sixth category was later added. These are:
  1. Healthy person.
  2. Mild systemic disease.
  3. Severe systemic disease.
  4. Severe systemic disease that is a constant threat to life.
  5. A moribund person who is not expected to survive without the operation.
  6. A declared brain-dead person whose organs are being removed for donor purposes.
  Participants
    ASA 1 | 21 | 25 | 46
    ASA 2 | 540 | 542 | 1082
    ASA 3 | 868 | 849 | 1717
    ASA 4 | 64 | 74 | 138

OUTCOME MEASURES:

1. Primary Outcome: Disability-free Survival
Description: Disability-free survival up to 1 year: survival and freedom from disability. The latter is defined as a persistent (≥6 months) reduction in health status as measured by a 12-item version (12-60 points) of World Health Organisation Disability Assessment Schedule score (WHODAS) of 24 points, reflecting a disability level of at least 25% and being the threshold point between "disabled" and "not disabled" as per WHO guidelines. Disability will be assessed by the participant, but if unable then we will use the proxy's report. The date of onset of new disability will be recorded. Further details are provided in the Procedures Manual and the Statistical Analysis Plan.
Time Frame: 1 year postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1493 | 1490
Participants | 165 | 172

2. Secondary Outcome: Death
Description: deceased within 12 months
Time Frame: 90 days, then up to 12 months after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1493 | 1490
Participants | 96 | 95

3. Secondary Outcome: Composite Septic Outcome or Death
Description: composite of 1 or more of:sepsis, surgical site infection, anastomotic leak, death and pneumonia
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1493 | 1490
Participants | 295 | 323

4. Secondary Outcome: Sepsis
Description: using Centers for Disease Control and Prevention (CDC) with National Healthcare Safety Network (NHSN) criteria, two or more features of the systematic inflammatory response syndrome (SIRS) plus evidence of a source or site of infection (can be positive blood culture or purulence from any site)
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1487 | 1481
Participants | 129 | 157

5. Secondary Outcome: Surgical Site Infection
Description: using CDC criteria (http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf):
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1481 | 1487
Participants | 245 | 202

6. Secondary Outcome: Pneumonia
Description: The presence of new and/or progressive pulmonary infiltrates on chest radiograph plus two or more of the following:
  1. Fever ≥ 38.5°C or postoperative hypothermia <36°C
  2. Leukocytosis ≥ 12,000 WBC/mm3 or leukopenia < 4,000 WBC/mm3
  3. Purulent sputum and/or
  4. New onset or worsening cough or dyspnoea.
Time Frame: 30 Days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1481 | 1487
Participants | 54 | 57

7. Secondary Outcome: Acute Kidney Injury
Description: according to The Kidney Disease: Improving Global Outcomes (KDIGO) group criteria, but not urine output - for Stage 2 or worse AKI defined as at least 2-fold increase in creatinine, or estimated GFR decrease >50%.(73) We also plan to report renal replacement therapy up to 90 days after surgery. Because a restrictive IV fluid regimen may artificially elevate serum creatinine due to a smaller dilutional effect from less IV fluids, we therefore calculated adjusted creatinine by first estimating the volume of distribution for creatinine as equal to total body water (assumed to be 60% of body weight, expressed in mL).
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1439 | 1443
Participants | 72 | 124

8. Secondary Outcome: Pulmonary Oedema
Description: respiratory distress or impaired oxygenation AND radiological evidence of pulmonary oedema
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1487 | 1481
Participants | 32 | 20

9. Secondary Outcome: Total Duration of Time Spend in the ICU or HDU (in Days)
Description: including initial ICU admission and readmission times up to 30 days post operatively
Time Frame: 30 day postoperative
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1493 | 1490
days | 1.8 [1.0 to 3.1] | 1.4 [0.9 to 2.9]

10. Secondary Outcome: Hospital Stay
Description: from the start (date, time) of surgery until actual hospital discharge
Time Frame: 30 days postoperative
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1493 | 1490
days | 5.6 [3.6 to 10.5] | 6.4 [3.6 to 10.6]

11. Secondary Outcome: Quality of Recovery
Description: 15-item Quality of Recovery Score. The score is a patient reported outcome measure to score the individuals recovery following anaesthesia and surgery. Minimum value is 0 and maximum value is 150. The score of 150 is good. The higher the score the better
Time Frame: days 3
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1418 | 1420
score on a scale | 107 [90 to 122] | 106 [89 to 121]

12. Secondary Outcome: Anastomotic Leak
Description: A defect of the intestinal wall at the anastomotic site (including suture and staple lines of neorectal reservoirs) leading to a communication between the intra- an extra luminal compartments.
Time Frame: 30 days postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1487 | 1481
Participants | 35 | 49

13. Secondary Outcome: C-reactive Protein
Description: plasma C-reactive protein (CRP, using site-specific assay) concentration on Day 3
Time Frame: Day 3 postoperative
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 1073 | 1068
mg/L | 133 [80 to 200] | 136 [82 to 198]

14. Secondary Outcome: mmol/L
Description: peak serum lactate within 24 hours of surgery
Time Frame: 24 hours post surgery
Measure: Median (Inter-Quartile Range); unit: mmol/L
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 436 | 404
mmol/L | 1.6 [1.1 to 2.4] | 1.6 [1.1 to 2.4]

15. Secondary Outcome: Total ICU Stay and Unplanned ICU Admission to ICU
Description: additive, including initial ICU admission and readmission times up to Day 30
Time Frame: 30 days postoperative
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Liberal | Restrictive
Number analyzed (Participants) | 473 | 485
days | 1.4 [0.9 to 2.9] | 1.8 [1.0 to 3.1]

16. Other Pre Specified Outcome: Preplanned Substudies (for Mechanistic Understanding)
Description: We plan several substudies (to be funded from other sources), each of which will have a separate protocol and authorship plan (using an expanded list of contributors). Additional blood tests and other investigations will be done at selected hospitals according to local interest and expertise.
  1. Cost-effectiveness, to include hospital stay and complications as we have done previously
  2. Hyperchloraemic acidosis (to measure strong ion difference, Cl-, lactate, albumin …)
  3. Pulmonary oedema and acute lung injury (to measure FiO2/PaO2 ratio, CT/CXR-confirmed atelectasis …)
  4. Perioperative oliguria and acute kidney injury 5. Obesity and perioperative risk 6. BNP and risk prediction 7. Goal directed therapy - decision analysis 8. Perioperative diabetes and HbA1C 9. CKD follow-up
Time Frame: 5 years
Reporting Status: Not Posted, anticipated posting 2026-11

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 30 days following surgery
Description: Please note that the patients reviewed for adverse events are the patients that completed the 30 day follow up data collection. There fore as per the Figure one according to follow up
Arm/Group | Liberal | Restrictive
All-Cause Mortality (participants affected / at risk) | 96/1493 | 95/1490
Serious Adverse Events (participants affected / at risk) | 295/1493 | 323/1490
Other Adverse Events (participants affected / at risk) | 78/1493 | 79/1490
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal (N=1493) | Restrictive (N=1490)
Surgical site infection (Infections and infestations) | 295 (295) | 323 (323) — Surgical site infection: using CDC criteria (http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf):
Sepsis (Infections and infestations) | 129 (129) | 157 (157) — Sepsis: using Centers for Disease Control and revention (CDC) with National Healthcare Safety Network (NHSN) criteria -two or more features of the systematic inflammatory response syndrome (SIRS) plus evidence of a source or site of infection.:
Anastomotic leak (Infections and infestations) | 35 (35) | 49 (49) — A defect of the intestinal wall at the anastomotic site (including suture and staple lines of neorectal reservoirs) leading to a communication between the intra- an extra luminal compartments
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 57 (57) | 54 (54)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liberal (N=1493) | Restrictive (N=1490)
Cardiovascular (Cardiac disorders) | 78 (78) | 79 (79)
Thrombolism (Blood and lymphatic system disorders) | 23 (23) | 31 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2016-08-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT01424150/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-29): https://cdn.clinicaltrials.gov/large-docs/50/NCT01424150/SAP_001.pdf